CLINICAL TRIAL: NCT04127240
Title: The Effect of Meat Intake as a Part of the DASH Diet on Indices of Muscular Fitness, Body Composition and Metabolic Health in Adults 65 and Older: A Controlled-Feeding Systems-Biology Study
Brief Title: The Effect of the DASH Diet Containing Meat on Muscle and Metabolic Health in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Dakota State University (Other)
Responsible Party: Principal Investigator, Cydne Perry, Assistant Professor, South Dakota State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1712006
Record Dates: First submitted 2019-10-10; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Obesity; Sarcopenia; Aging
MeSH Terms: conditions — Obesity; Sarcopenia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meat assignment in DASH intervention (Experimental): Participants consumed 3 ounces of red meat per day as a part of the DASH diet.
  Interventions: Other: DASH diet containing daily intakes of red meat
- Meat allocation in DASH intervention (Experimental): Participants consumed 6 ounces of red meat per day as a part of the DASH diet.
  Interventions: Other: DASH diet containing daily intakes of red meat

INTERVENTIONS:
Other: DASH diet containing daily intakes of red meat — Each participant was randomized to consume 3 or 6 ounces of red meat as a part of the DASH dietary pattern for 12-weeks.

SUMMARY:
Age-related changes in body composition, muscular fitness, and metabolic health resulting in the onset of obesity, sarcopenia, and chronic diseases are profound public health issues that are in need of immediate attention. Effective and feasible methods, such as dietary therapies, are needed to improve health in older adults that in turn lead to independence, enhanced quality of life and reduced hospitalizations. Diet quality and dietary protein intake are vital for maintaining body composition, muscle mass and improved physical performance. Malnutrition in dietary protein intake is a major cause of reduced muscle mass, strength, and function in older adults. The Dietary Approaches to Stop Hypertension (DASH) dietary pattern is a high-quality therapeutic diet known to improve health status in various diverse and at-risk populations resulting in improved heart health, maintained cognitive function and reductions in metabolic diseases such as diabetes, metabolic syndrome, and nonalcoholic fatty liver disease. The primary protein recommendations of the DASH diet are poultry and fish and it is recommended to decrease or exclude red meats from the diet. However, studies have demonstrated that lean red meat incorporated into a DASH-like diet doesn't exacerbate cardiovascular health indices in adults, indicating that lean red meat can be included in the DASH diet without negative effects on heart health. Although studies have reported on the DASH diet in older adults, no studies have investigated the effect of the DASH diet containing lean red meat on measures of body composition, muscle mass or metabolic health under controlled-feeding conditions. The purpose of this study was to determine the effect of the DASH diet containing daily intakes of lean red meat on indicators of body composition, muscular fitness and biomarkers of metabolic health in adults 65 and older using controlled-feeding and systems biology approaches.

ELIGIBILITY:
Inclusion Criteria:

* 65 and older
* Upward mobile ability

Exclusion Criteria:

* Under the age of 65
* Immobility

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-11-10 (Actual); Study Completion 2018-11-10 (Actual)

PRIMARY OUTCOMES:
Body weight | Change in body weight from baseline to 3 months
  Measured by bioelectrical impedance
Hand grip strength | Change in strength from baseline to 3 months
  Measured by a hand-held dynamometer
Glucose | Change in glucose concentrations from baseline to 3 months
  Measure serum glucose using colorimetry assay

CONTACTS AND LOCATIONS:
Overall Officials: Cydne A Perry, PhD, Principal Investigator — South Dakota State University
Locations (1):
- South Dakota State University, Brookings, South Dakota, United States

REFERENCES:
- [Derived] Perry CA, Van Guilder GP, Butterick TA. Decreased myostatin in response to a controlled DASH diet is associated with improved body composition and cardiometabolic biomarkers in older adults: results from a controlled-feeding diet intervention study. BMC Nutr. 2022 Mar 15;8(1):24. doi: 10.1186/s40795-022-00516-9. PMID 35287731